CLINICAL TRIAL: NCT06622733
Title: Attitude Towards the Concept of Cesarean Section on Demand Among a Random Sample of Pregnant Women Attending the Antenatal Care Clinic of Sohag University Hospital
Brief Title: Attitude Towards the Concept of CS on Demand
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Khalifa Mohamed, Residence at gyn and OBS department, Sohag University
Other Study IDs: Soh-Med-24-09---12MS
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Cs
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Questionnaire — Attitude towards the concept of CS on demand

SUMMARY:
Caesarean section (CS) is a surgical procedure performed to facilitate delivery of the baby through an incision made on the mother's abdomen. Ideally, it is recommended in situations where normal vaginal delivery (VD) can pose risks to either the mother baby or both . In the western world women have only one or two children, while in the East or the Middle East, women are culturally coerced into having many children. Thus, they are more prone to multiple Cesarean deliveries in their lifetime [1.2]. ThisAccording to the World Health Organization (WHO), since 1985, the acceptable percentage of worldwide C-sections has been 10-15% of all deliveries [3]. One of the most critical findings of the American Center for Disease Control and Prevention found that the Cesarean delivery rate has increased from 20.7% in 1995 to 31.6% in 2016 [4 ]. It is important to mention that Cesarean deliveries are life-saving procedures when there are obstetrical indications.(5.6) Cesarean delivery indications include fetal malpresentation, multiple pregnancies, chorioamnionitis, arrested labour, oligohydramnios, cord prolapse, cephalo-pelvic disorders, and medical diseases such as eclampsia and HELPP (hemolysis, elevated liver enzymes, and low platelets) syndrome .the number of patients undergoing Cesarean delivery for non-obstetric reasons has rapidly increased. This could be due to many factors influencing the patients' decisions, including possible fetal outcomes concerning beliefs in some cultures and the convenience of patients and obstetricians(7) .cesarean section on demand allows a woman to choose a cesarean section without a medical reason, based solely on her personal preference Five themes that reflected the reasons for elective cesarian birth without medical indication were identified: (1) fear of vaginal birth process, (2) concerns about future sexual life, (3) need for humanized birth, (4) personal reasons, and (5) decision-making process.(8) raising the awareness of providers about the appropriate indications for CS and the importance of advocating for vaginal delivery among eligible women - including those with a previous CScan trigger practice changes that may reduce the incidence of non-medically indicated caesarean delivery

ELIGIBILITY:
Inclusion Criteria:

* pregnant women attending the antenatal care clinic of Sohag University hospital

Exclusion Criteria:

* postmenopausal women
* women with previous two or more cs
* women refusing to participate in the questionnaire

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women attending the antenatal care clinic of Sohag University hospital
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-09-28 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Women's interest in caesarean section | 6 months
  Questionnaire to inform women about benefits and risks of CS

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sobande A, Eskandar M. Multiple repeat caesarean sections: complications and outcomes. J Obstet Gynaecol Can. 2006 Mar;28(3):193-197. doi: 10.1016/S1701-2163(16)32105-3. PMID 16650356
- [Background] Betran AP, Torloni MR, Zhang JJ, Gulmezoglu AM; WHO Working Group on Caesarean Section. WHO Statement on Caesarean Section Rates. BJOG. 2016 Apr;123(5):667-70. doi: 10.1111/1471-0528.13526. Epub 2015 Jul 22. No abstract available. PMID 26681211
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Kirmeyer S, Mathews TJ, Wilson EC. Births: final data for 2009. Natl Vital Stat Rep. 2011 Nov 3;60(1):1-70. PMID 22670489
- [Background] Abbaspoor Z, Moghaddam-Banaem L, Ahmadi F, Kazemnejad A. Iranian mothers' selection of a birth method in the context of perceived norms: a content analysis study. Midwifery. 2014 Jul;30(7):804-9. doi: 10.1016/j.midw.2013.06.003. Epub 2013 Jul 17. PMID 23870747